CLINICAL TRIAL: NCT06151184
Title: The Effects of Chiropractic Manual Adjustments on Nervous System Function in Individuals with Post-concussion Syndrome: a Proof of Concept Trial
Brief Title: Post-concussion Syndrome and Chiropractic
Acronym: PCS
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Life University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: I-0025
Record Dates: First submitted 2023-11-21; First posted 2023-11-30 (Actual); Last update posted 2025-02-12 (Actual); Status verified 2025-02

CONDITIONS: Post-Concussion Syndrome
Keywords: chiropractic care; spinal manipulation; heart rate variability; autonomic nervous system; electroencephalography; interlimb symmetry; impedance cardiography; electrocardiography; electrodermal activity; chiropractic adjustment; chiropractic
MeSH Terms: conditions — Post-Concussion Syndrome | interventions — Manipulation, Chiropractic

STUDY DESIGN:
Intervention Model Description: The intervention for this proof-of-concept trial is chiropractic manual adjustments. Participants will undergo chiropractic care from a state licensed chiropractor. Each individual's care plan will be determined by that individual and their specific field doctor for frequency of visits and type of chiropractic technique used. Participants will undergo 6 weeks of chiropractic for this study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Post-concussion syndrome participants (Experimental): Post-concussion syndrome participants will all receive manual chiropractic adjustment interventions.
  Interventions: Procedure: Chiropractic adjustment

INTERVENTIONS:
Procedure: Chiropractic adjustment — 6 weeks of chiropractic care, with frequency and type of procedures determined by field clinician after initial examination.

SUMMARY:
This proof-of-concept trial will explore the effects of manual chiropractic adjustments on nervous system function in individuals with post-concussion syndrome. This study will aim to recruit 10 individuals to receive 6 weeks of chiropractic care with 3 assessment periods. The participants will undergo a baseline assessment, mid-trial assessment, and post-trial assessment. The participants will wear an electroencephalography (EEG) cap for a neural assessment during an event related potential. They will wear electrical diodes to measure electrocardiography (ECG), impedance cardiography (ICG), and electrodermal activity (EDA) throughout the study and during an orthostatic challenge. Additional sensors will be placed on the participant to measure interlimb symmetry patterns during gait while walking on a treadmill.

DETAILED DESCRIPTION:
Participants enrolled in the study will take a screening questionnaire to first determine eligibility. Once qualified, each individual will undergo a physical exam by a state licensed chiropractor to determine if there are any contraindications to undergo chiropractic care throughout the duration of the study. Each participant will receive 6 weeks of chiropractic care and will be assessed at weeks 0, 2, and 6 at the Dr. Sid E Williams Center for Chiropractic Research. Each participant will perform a number of tests to determine the evaluated function of their nervous system. In total, 3 different tests will be performed by the participant during an assessment visit that will take approximately 2.5 - 3 hours. During the assessments, each individual will be wearing electrical diodes to continually monitor ECG, ICG, and EDA. The specific assessments will be as follows:

1. Wearing an EEG net and then perform an event related potential after a baseline recording
2. Performing an orthostatic challenge while measuring ECG, ICG, and EDA
3. Wearing motion sensors while walking at a comfortable pace on a treadmill to evaluate interlimb symmetry and gait dynamics

ELIGIBILITY:
Inclusion Criteria:

* 18 or older
* Diagnosed by a physician with post-concussion syndrome OR self-identifies as having a concussion based on responses to the HELPS screening tool
* Has at least 3 of the following chronic symptoms at least 3 months since concussion: headache; dizziness; insomnia; fatigue; concentration difficulty; memory difficulty; intolerance to stress, emotions, and alcohol; irritability
* Able to understand and communicate in English
* Able to make informed decisions without assistance
* Can wear an EEG net for 40 minutes
* Can sit quietly for at least 15 minutes
* Capable of walking on a treadmill at a comfortable pace for 10 minutes consecutively
* Capable of moving from a supine to standing to supine position quickly and safely
* Able to wear multiple electrodes placed on chest, back, and fingertips
* Able to wear multiple sensors placed on head, back, pelvis, hands, arms, and legs
* Has not had a chiropractic adjustment within the last one month
* Has not received any other interventions within the past one month such as osteopathic spinal manipulation, physical therapy rehabilitation or manipulation, massage, body movement therapies, or acupuncture

Exclusion Criteria:

* Diagnosed with a serious mental disorder such as schizophrenia or bipolar disorder
* Has malignant hypertension, which is a condition whereby their blood pressure rises suddenly and quickly
* Has a known condition that causes syncope with postural changes, such as POTS
* Has an implanted device (i.e., pacemaker)
* Has a physical disability affecting their gait
* Has a history of previous surgery or injury to the musculoskeletal structures or skull in the past three months
* Has a prosthetic for any extremity
* Has a hearing impairment or uses a hearing aid
* History of stroke
* Taking short-acting benzodiazepines, which includes midazolam and triazolam
* Involved with current litigation related to a physical health-related injury
* Untreated diagnosed osteoporosis or articular instability such as atlanto-axial instability
* Currently pregnant
* Unwilling to wash hair/head and remove hair products, accessories, braids, or wigs for assessment appointments
* Deemed high-risk using the Columbia-Suicide Severity Rating Scale (C-SSRS) and referred for further evaluation (assessed at initial session in lab)
* Experiences daily/chronic pain >3 out of 10 on the visual analog scale (VAS)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2024-01-27 (Actual); Primary Completion 2026-03 (Estimated); Study Completion 2026-07-31 (Estimated)

PRIMARY OUTCOMES:
Participant recruitment | 24 months (recruitment period)
  Average number of participants recruited/enrolled per month
Participant scheduling | 24 months (recruitment period)
  Average time lag between first lab assessment & first chiropractic visit
Participant compliance | 24 months (recruitment period)
  % of participants violating 1 or more pre-assessment lifestyle restrictions & unable/unwilling to be rescheduled
Participant adherence | 24 months (recruitment period)
  % of participants not attending ≥80% of their chiropractic sessions
Participant tolerability | 24 months (recruitment period)
  % of participants unable/unwilling to complete a given assessment
Participant retention | 24 months (recruitment period)
  % of participants completing the trial
Assessment acceptability | 24 months (recruitment period)
  Most common participant-rated acceptability score for each assessment process/procedure
Intervention acceptability | 24 months (recruitment period)
  Most common participant-rated acceptability score for each aspect of the chiropractic care
Data fidelity | 24 months (recruitment period)
  % of acquisitions from a given assessment that are unsuitable for analysis
Implementation acceptability | 24 months (recruitment period)
  Most common clinician-rated acceptability score for each trial process/procedure

SECONDARY OUTCOMES:
EEG resting state broadband power | Day 1
  64-channel hydronet cap
EEG resting state broadband power | Week 2
  64-channel hydronet cap
EEG resting state broadband power | Week 6
  64-channel hydronet cap
EEG resting state functional connectivity | Day 1
  64-channel hydronet cap
EEG resting state functional connectivity | Week 2
  64-channel hydronet cap
EEG resting state functional connectivity | Week 6
  64-channel hydronet cap
EEG evoked latency | Day 1
  64-channel hydronet cap during auditory oddball task
EEG evoked latency | Week 2
  64-channel hydronet cap during auditory oddball task
EEG evoked latency | Week 6
  64-channel hydronet cap during auditory oddball task
ECG mean interbeat interval | Day 1
  3 sensors on torso
ECG mean interbeat interval | Week 2
  3 sensors on torso
ECG mean interbeat interval | Week 6
  3 sensors on torso
ECG respiratory sinus arrhythmia (RSA) | Day 1
  3 sensors on torso
ECG respiratory sinus arrhythmia (RSA) | Week 2
  3 sensors on torso
ECG respiratory sinus arrhythmia (RSA) | Week 6
  3 sensors on torso
ECG de-trended fluctuation analysis | Day 1
  3 sensors on torso
ECG de-trended fluctuation analysis | Week 2
  3 sensors on torso
ECG de-trended fluctuation analysis | Week 6
  3 sensors on torso
Impedance cardiogram (ICG) pre-ejection period (PEP) | Day 1
  2 sensors on chest and 2 sensors on back
Impedance cardiogram (ICG) pre-ejection period (PEP) | Week 2
  2 sensors on chest and 2 sensors on back
Impedance cardiogram (ICG) pre-ejection period (PEP) | Week 6
  2 sensors on chest and 2 sensors on back
Impedance cardiogram (ICG) initial systolic time interval (ISTI) | Day 1
  2 sensors on chest and 2 sensors on back
Impedance cardiogram (ICG) initial systolic time interval (ISTI) | Week 2
  2 sensors on chest and 2 sensors on back
Impedance cardiogram (ICG) initial systolic time interval (ISTI) | Week 6
  2 sensors on chest and 2 sensors on back
Electrodermal activity (EDA) non-specific skin conductance responses (SCR) | Day 1
  2 sensors on first and second digits of non-dominant hand
Electrodermal activity (EDA) non-specific skin conductance responses (SCR) | Week 2
  2 sensors on first and second digits of non-dominant hand
Electrodermal activity (EDA) non-specific skin conductance responses (SCR) | Week 6
  2 sensors on first and second digits of non-dominant hand
Electrodermal activity (EDA) skin conductance level (SCL) | Day 1
  2 sensors on first and second digits of non-dominant hand
Electrodermal activity (EDA) skin conductance level (SCL) | Week 2
  2 sensors on first and second digits of non-dominant hand
Electrodermal activity (EDA) skin conductance level (SCL) | Week 6
  2 sensors on first and second digits of non-dominant hand
Composite Autonomic Symptom Score (COMPASS-31) | Day 1
  31-item questionnaire
Composite Autonomic Symptom Score (COMPASS-31) | Week 2
  31-item questionnaire
Composite Autonomic Symptom Score (COMPASS-31) | Week 6
  31-item questionnaire
Patient-Reported Outcomes Measurement Information System (PROMIS-29) | Day 1
  29-item questionnaire
Patient-Reported Outcomes Measurement Information System (PROMIS-29) | Week 2
  29-item questionnaire
Patient-Reported Outcomes Measurement Information System (PROMIS-29) | Week 6
  29-item questionnaire
Patient-Reported Outcomes Measurement Information System Cognitive Abilities and Cognitive Concerns Scale (PROMIS-Cog-8) | Day 1
  8-item questionnaire
Patient-Reported Outcomes Measurement Information System Cognitive Abilities and Cognitive Concerns Scale (PROMIS-Cog-8) | Week 2
  8-item questionnaire
Patient-Reported Outcomes Measurement Information System Cognitive Abilities and Cognitive Concerns Scale (PROMIS-Cog-8) | Week 6
  8-item questionnaire
Perceived Stress Scale (PSS) | Day 1
  10-item questionnaire
Perceived Stress Scale (PSS) | Week 2
  10-item questionnaire
Perceived Stress Scale (PSS) | Week 6
  10-item questionnaire
Post-Concussion Symptom Scale | Day 1
  22-item questionnaire
Post-Concussion Symptom Scale | Week 2
  22-item questionnaire
Post-Concussion Symptom Scale | Week 6
  22-item questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Ahmed Qazi, Principal Investigator — Life University
Locations (1):
- Dr. Sid E. Williams Center for Chiropractic Research, Marietta, Georgia, United States

IPD SHARING:
Plan to Share IPD: No